CLINICAL TRIAL: NCT04889131
Title: Yoga for Seniors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 vulnerable participant population
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Bader Philanthropies (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-0479; A176000 (Other: UW Madison); EDUC/KINESIOLOGY (Other: UW Madison)
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Aging Well
Keywords: Yoga; social isolation; underserved populations; elderly; movement; activity
MeSH Terms: conditions — Social Isolation; Motor Activity | interventions — Fitness Trackers

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to immediately begin a 12-week yoga class or complete a 12-week wait (wait-list control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Program (Experimental): 12-week yoga program begins immediately
  Interventions: Behavioral: Yoga Program Immediately; Other: Activity Monitor
- Wait-list Control (Active Comparator): Wait-listed to take the Yoga Program in 12-weeks time
  Interventions: Behavioral: Wait-Listed Control; Other: Activity Monitor

INTERVENTIONS:
Behavioral: Yoga Program Immediately — free 12 week yoga program, twice a week for 75 minutes each
  Arms: Yoga Program
Behavioral: Wait-Listed Control — assigned to take the Yoga Program in 12-weeks
  Arms: Wait-list Control
Other: Activity Monitor — Garmin VivoSmart activity monitor throughout study

SUMMARY:
The overall purpose of this study is to deliver a 12-week yoga program to older adults (over 60 years of age) in rural WI who do not have access to yoga programming and examine the effects of the programming on activities of daily living, gait, balance, falls, activity level and social isolation.

DETAILED DESCRIPTION:
Participants will be assigned to immediately begin a 12-week yoga class (2 classes per week for 75 minutes each) or complete a 12-week wait (wait-list control). The measures of interest will be examined at pretest (wait-list only), baseline, posttest and at 3-month follow-up to see what, if any, changes are maintained after completion of the program. All assessment data collections sessions will be conducted on-site at a predetermined site identified by the community partners.

ELIGIBILITY:
Inclusion Criteria:

* Ability to independently ambulate for at least 10 minutes continuously (with or without an assistive device)
* Ability to attend the yoga class for all or most of the 12 weeks
* A previous fall, near-fall or identified fear of falling

Exclusion Criteria:

* No known contraindication for exercise (i.e. a medical doctor has told you not to exercise)
* A resent injury that causes pain during movement
* Current enrollment in another research study or class focused on balance

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Change in MiniBESTest Score | [pre-test for waitlist group 3 months prior to class], baseline, post-test (3-months), 3-month follow up (6-months)
  The mini-BESTest will be used to assess balance. This 14-item, clinical battery is used to assess balance in four component areas (anticipatory transitions, postural response, sensory orientation and dynamic gait) and provides a single number summary of balance performance. Scores range from 0 to 28, with higher scores indicating higher function.
Change in Fall Frequency | [pre-test for waitlist group 3 months prior to class], baseline, post-test (3-months), 3-month follow up (6-months)
  Change in the frequency of falls will be assessed using a forced-choice paradigm: none, once, 2 to 10 times, weekly, or daily over the last 6 months.
Change in the Canadian Occupational Performance Measures (COPM) | [pre-test for waitlist group 3 months prior to class], baseline, post-test (3-months), 3-month follow up (6-months)
  The COPM is composed of the following steps: 1) participant identifies occupational performance problems for self-care and productivity, 2) participant rates each issue on a score of 1-10 (higher scores are more important), 3) participant chooses 5 most important problems, 4) participant rates each issue (1-10) for performance and satisfaction, 5) average score for each (performance and satisfaction) are calculated. Final score for each is 1-10 with higher scores better.
Change in Activities-Specific Balance Confidence Scale (ABC) | [pre-test for waitlist group 3 months prior to class], baseline, post-test (3-months), 3-month follow up (6-months)
  The ABC Scale measures a fear of falling. It is a 16-item survey where participants rate their level of self-confidence (0-100, where 100 is the highest self-confidence) for each item. The average score is reported.

SECONDARY OUTCOMES:
Change in Standardized Gait Analysis: Gait Velocity | [pre-test for waitlist group 3 months prior to class], baseline, post-test (3-months), 3-month follow up (6-months)
  Using the GaitRite® System, the temporal and spatial parameters of each participant will be captured during walking. The GaitRite® mat is a 14 foot portable electronic walkway, embedded with sensors to enable the measurement spatiotemporal variables of gait such as cadence, normalized velocity, stride length, base of support, and percent of cycle in double support. Participants will begin at a starting point two meters from the mat, then walk toward and step onto the mat to continue walking until they achieve the stop line located two meters off of the opposite side of the mat. Data will be collected for forward preferred speed, backward preferred speed, forward fast, tandem and dual task gait. Each participant will complete five trials for each condition.

OTHER OUTCOMES:
Change in Activity Level Measured by Number of Steps Taken | [pre-test for waitlist group 3 months prior to class], baseline, post-test (3-months), 3-month follow up (6-months)
  Participants will be fitted with a Garmin VivoSmart activity monitor and will be asked to wear the device for the duration of the study.
Change in Performance Assessment of Self-Care Skills (PASS) | [pre-test for waitlist group 3 months prior to class], baseline, post-test (3-months), 3-month follow up (6-months)
  The Performance Assessment of Self-Care Skills (PASS) assesses basic self-care and instrumental activities of daily living. Subscales: Independence, Safety, and Adequacy (0-3 where higher scores indicate less difficulty with basic self-care).

CONTACTS AND LOCATIONS:
Overall Officials: Kristen A Pickett, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No